CLINICAL TRIAL: NCT06037551
Title: Evaluierung Des Blutglukose Monitoring Systems Contour Care Der Firma Ascensia Diabetes Care Deutschland GmbH gemäß DIN EN ISO 15197:2015
Brief Title: System Accuracy of the Blood Glucose Monitor for Personal Use Contour Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut fur Diabetes Karlsburg GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023_005
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subject glucometer measurement (Experimental): Blood glucose measurement BGM for personal use
  Interventions: Diagnostic Test: blood glucose measuremen subject; Diagnostic Test: blood glucose measuremen reference
- glucometer measurement (Experimental): evaluation of repeatability measurement precision
  Interventions: Diagnostic Test: blood glucose measuremen reference

INTERVENTIONS:
Diagnostic Test: blood glucose measuremen subject — measurement of the blood glucose concentration of subject using BGM and capillary finger tip blood
  Arms: Subject glucometer measurement
Diagnostic Test: blood glucose measuremen reference — measurement of the blood glucose concentration of subject using reference method and capillary finger tip blood

SUMMARY:
This study assesses the system accuracy of a blood glucose monitoring system in accordance with DIN EN ISO 15197:2015

ELIGIBILITY:
Inclusion criteria:

* Male or female patients with hypo-, eu- or hyperglycaemia
* The written informed consent had to be signed
* The volunteers must be older than 18 years
* The volunteers have legal capacity and are able to understand meaning, nature and possible consequences of the procedures involved

Exclusion criteria:

* Pregnancy or lactation
* Acute or chronic diseases with the risk of aggravation by the measure
* A current constitution that does not allow participating in the study
* Participation in another study or activity with the blood glucose measuring system evaluated in the present study
* Application of substances listed in Appendix A of DIN EN ISO 15197:2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Analysis of system accuracy based on DIN EN ISO 15197 | 1 Day
  Assessment of the analytical measurement performance of the blood glucose monitor based on procedures defined in DIN EN ISO 15197

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Rebrin, PhD, Study Director — Institut fur Diabetes Karlsburg GmbH
Locations (1):
- Institut für Diabetes Karlsburg GmbH, Karlsburg, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: Undecided
optional: age, blood glucose levels and hematocrit of subjects